CLINICAL TRIAL: NCT07120945
Title: A Prospective, Multicenter, Single-arm Pre-market Study of the Medtronic Hugo™ Robotic-Assisted Surgery (RAS) System in Gynecological Subjects (Embrace Gynecology)
Brief Title: Hugo™ Robotic-Assisted Surgery (RAS) System in Gynecological Subjects (Embrace Gynecology)
Acronym: Embrace Gyn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT24040
Record Dates: First submitted 2025-07-31; First posted 2025-08-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Uterine Fibroids (UF); Menstrual Disorders; Adenomyosis of Uterus; Endometriosis; Uterine Prolapse; Precancerous/Nonmalignant Condition; Cervical Cancer; Endometrial Cancer; Ovarian Cancer
MeSH Terms: conditions — Leiomyoma; Menstruation Disturbances; Adenomyosis; Endometriosis; Uterine Prolapse; Precancerous Conditions; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms | interventions — Robotic Surgical Procedures; Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Robotic-Assisted Surgery (RAS) Hysterectomy Procedures (Experimental): Patients indicated for Robotic-Assisted Surgery (RAS) for hysterectomy procedures (radical, modified radical, or total hysterectomy), inclusive of subjects being treated for malignancies.
  Interventions: Device: Robotic Assisted-Surgery (RAS) Hysterectomy

INTERVENTIONS:
Device: Robotic Assisted-Surgery (RAS) Hysterectomy — Patients indicated for Robotic Assisted-Surgery (RAS) hysterectomy procedures will have the RAS surgery using the Medtronic Hugo™ RAS system.

SUMMARY:
The purpose of this research is to evaluate the safety and performance of the investigational Medtronic Hugo™ Robotic Assisted Surgery (RAS) system when used during hysterectomy procedures, including patients being treated for cancer.

DETAILED DESCRIPTION:
This study will enroll up to 70 subjects and conducted using up to five investigational sites in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 22 years) as required by local law
2. Patients indicated for a hysterectomy (radical, modified radical, or total hysterectomy) inclusive of subjects being treated for malignancies with the Hugo™ RAS system
3. Patient is an acceptable candidate for a fully robotic-assisted surgical procedure, a laparoscopic surgical procedure, and an open surgical procedure
4. The patient is willing to participate and consents to participate, as documented by a signed and dated informed consent form

Exclusion Criteria:

1. Patient for whom minimally invasive surgery is contraindicated as determined by the Investigator.
2. Patients with comorbidities or medical characteristics which would preclude the surgical procedure in the opinion of the Investigator.
3. Patients with an estimated life expectancy of less than 6 months as determined by Investigator
4. Patients diagnosed with a bleeding disorder and/or who cannot be removed from their anticoagulants prior to surgery based on surgeon discretion and standard-of-care
5. Patients who are pregnant at the time of the surgical procedure.
6. Patients who are considered to be part of a vulnerable population (e.g., prisoners or those without sufficient mental capacity).
7. Patients who have participated or are currently participating in an investigational drug or in a device research study that may interfere with this study in the opinion of the Investigator.
8. Patients with active infections including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia at physicians' discretion.
9. Patients with a pre-surgical diagnosis of recurring cancer and gross metastatic conditions are excluded.

   I. For cervical cancer, only patients with Stages 1a1, 1a2, 1b1, may be included, and within these stages, II. Eligibility is further restricted to those with Stage IB1 tumors less than 2 cm (on MRI) and less than 10 mm stromal invasion on excisional biopsy, or less than 50% cervical stromal invasion (on MRI).

   III. All other cervical cancer stages are excluded from the study.
10. Patients with disease spread out of the pelvis requiring surgical intervention with surgical expertise outside of the gynecological space, with the exception of para-aortic lymph node dissection, as determined by the investigator.
11. Patients who have a body mass index (BMI) > 44.1 kg/m2

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | Intraoperative
  Surgical success rate is the procedure utilizing Hugo™ as outlined in the preoperatively defined surgical plan without conversion to an alternative robotic-assisted system, laparoscopy, or open surgery.

SECONDARY OUTCOMES:
Operative time | Intraoperative
  Time from skin incision to skin closure
Hospital length of stay | From procedure to discharge, through approximately 30 days
  Hospital length of stay from the date of the procedure to discharge
Major complication rate | 30 Days
  Overall rate of subjects with one or more complication (Clavien-Dindo Grade III or higher) related to study device and/or procedure, from the first incision through 30 days post-procedure.
Complication rate | 30 Days
  Overall rate of subjects with one or more complications (Clavien-Dindo Grade I or higher) related to study device and/or procedure, from the first incision through 30 days post-procedure.
Rate of intraoperative adverse events | Intraoperative
  Rate of intraoperative adverse events related to study device and/or procedure from first incision through skin closure.
Rate of readmission | 30 Days
  Rate of readmission within 30 days due to device and/or procedure related adverse events.
Rate of therapy-specific adverse events | 3 Months
  Rate of complications due to the study device and/or procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Rossi, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Ascension St. Vincent's Riverside, Jacksonville, Florida
  - The University of South Florida, Tampa, Florida
  - Duke University, Durham, North Carolina
  - Allegheny Health Network - West Penn, Pittsburgh, Pennsylvania